CLINICAL TRIAL: NCT01912781
Title: Clinical Evaluation of the Safety and Efficacy of FID 120947A Compared to a Marketed Lens Care Solution in Gas Permeable Contact Lens Wearers
Brief Title: Safety and Efficacy Evaluation of a New Contact Lens Disinfecting Solution in Gas Permeable Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: C-13-004
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Myopia; Astigmatism; Hyperopia; Refractive Error
Keywords: contact lenses; contact lens solution; gas permeable contact lenses
MeSH Terms: conditions — Myopia; Astigmatism; Hyperopia; Refractive Errors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 120974A (Experimental): FID 120947A contact lens disinfecting solution used with gas permeable contact lenses (study lenses) on a daily basis for 90 days
  Interventions: Device: FID 120947A contact lens disinfecting solution; Device: Gas permeable contact lenses
- Boston Simplus (Active Comparator): Boston Simplus multi-action solution used with gas permeable contact lenses (study lenses) on a daily basis for 90 days
  Interventions: Device: Boston Simplus multi-action solution; Device: Gas permeable contact lenses

INTERVENTIONS:
Device: FID 120947A contact lens disinfecting solution — Investigational 3% hydrogen peroxide solution intended for simultaneous cleaning, protein removal, disinfecting and storage of gas permeable contact lenses
  Other Names: Clear Care® Plus
  Arms: FID 120974A
Device: Boston Simplus multi-action solution — Commercially available solution indicated for cleaning, removing protein, rinsing, disinfecting, conditioning, storing and cushioning of fluoro silicone acrylate and silicone acrylate rigid gas permeable contact lenses
  Arms: Boston Simplus
Device: Gas permeable contact lenses — Commercially available gas permeable contact lenses worn a minimum of 8 hours each day on a daily wear basis for the duration of the study (90 days).
  Other Names: Boston XO; Boston II

SUMMARY:
The purpose of this study is demonstrate substantial equivalence of an investigational contact lens disinfecting solution to a commercially available contact lens solution in gas permeable lens wearers.

DETAILED DESCRIPTION:
Subjects with normal eyes (other than correction for refractive error) successfully wearing silicone acrylate or fluoro silicone acrylate gas permeable contact lenses were randomized 2:1 to receive either the investigational or commercial contact lens solution for daily use throughout the study (90 days).

ELIGIBILITY:
Inclusion Criteria:

* Normal eyes (other than correction for visual acuity);
* Successful history of gas permeable contact lens wear in both eyes in one of two brands: Boston XO or Boston II;
* Best spectacle corrected distance visual acuity greater than or equal to 20/25 in each eye;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular or systemic medical condition that may, in the opinion of the investigator, preclude safe administration of the investigational products or affect the results of this study;
* Need to wear contact lenses on an extended wear basis (ie, overnight) during the study;
* Use of a daily cleaner and/or an enzyme cleaner to care for lenses at least 7 days prior to Visit 1;
* History of intolerance or hypersensitivity to any component of the investigational products;
* Use of all over-the-counter (OTC) or prescribed topical ocular medications within 7 days prior to Visit 1;
* Moderate, severe, abnormal, or other ocular findings;
* Current or history of ocular infection, severe inflammation, or disease within 6 months prior to Visit 1;
* Any systemic disease at Visit 1 (including allergies, respiratory infections or colds) that may affect the eye or be exacerbated by use of contact lenses or contact lens solutions;
* Use of systemic medications that may contribute to adverse ocular effects unless on a stable dosing regimen;
* Ocular surgery within the last 12 months;
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lieve Convents, Lead CSM, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 12 study centers located in the US.
Pre-assignment Details: Of the 112 enrolled, 2 subjects were exited as screen failures and 4 were discontinued prior to randomization. This reporting group includes all randomized subjects (106).
Groups:
- FID 120974A: Contact lens disinfecting solution used with gas permeable contact lenses (study lenses) on a daily basis for 90 days
- Boston Simplus: Multi-action solution used with gas permeable contact lenses (study lenses) on a daily basis for 90 days
Period: Overall Study
Arm/Group | FID 120974A | Boston Simplus
Started | 71 | 35
Completed | 69 | 35
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | FID 120974A | Boston Simplus | Total
Number analyzed (Participants) | 71 | 35 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (10.2) | 50.5 (13.4) | 52.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 28 | 83
  Male | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Visibly Clean Lenses
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered. A lens was considered visibly clean if it had nondetectable films or deposits. One eye (study eye) contributed to the analysis.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all subjects with data at visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 69 | 35
percentage of subjects
  Day 7 | 42.0 | 57.1
  Day 30 | 29.0 | 42.9
  Day 60 | 29.0 | 42.9
  Day 90 | 30.4 | 31.4

2. Primary Outcome: Percentage of Subjects With Crystalline Deposits by Type
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered: Type II = films or deposits visible only under special conditions, such as special illumination using an eyepiece of 7-10 times magnification, Type III = films or deposits readily visible on a dry lens under room lighting, with unaided eye, and Type IV = films or deposits obvious under room lighting, with unaided eye, when the lens is wet or dry. One eye (study eye) contributed to the analysis.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all randomized subjects. Here, "n" is the total number of subjects with crystalline deposits in each treatment group, respectively, by visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 71 | 35
percentage of subjects
  Day 7, Type II, n=10, 5 | 90.0 | 80.0
  Day 7, Type III, n=10, 5 | 0.0 | 20.0
  Day 7, Type IV, n=10, 5 | 10.0 | 0.0
  Day 30, Type II, n=17, 3 | 70.6 | 100.0
  Day 30, Type III, n=17, 3 | 17.6 | 0.0
  Day 30, Type IV, n=17, 3 | 11.8 | 0.0
  Day 60, Type II, n=18, 8 | 61.1 | 87.5
  Day 60, Type III, n=18, 8 | 16.7 | 0.0
  Day 60, Type IV, n=18, 8 | 22.2 | 12.5
  Day 90, Type II, n=21, 10 | 61.9 | 60.0
  Day 90, Type III, n=21, 10 | 23.8 | 10.0
  Day 90, Type IV, n=21, 10 | 14.3 | 30.0

3. Primary Outcome: Percentage of Subjects With Film Deposits by Type
Description: as for outcome 2
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all randomized subjects. Here, "n" is the total number of subjects with film deposits in each treatment group, respectively, by visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 71 | 35
percentage of subjects
  Day 7, Type II, n=40, 15 | 80.0 | 66.7
  Day 7, Type III, n=40, 15 | 7.5 | 26.7
  Day 7, Type IV, n=40, 15 | 12.5 | 6.7
  Day 30, Type II, n=47, 20 | 72.3 | 80.0
  Day 30, Type III, n=47, 20 | 10.6 | 10.0
  Day 30, Type IV, n=47, 20 | 17.0 | 10.0
  Day 60, Type II, n=47, 20 | 74.5 | 80.0
  Day 60, Type III, n=47, 20 | 21.3 | 5.0
  Day 60, Type IV, n=47, 20 | 4.3 | 15.0
  Day 90, Type II, n=45, 24 | 73.3 | 79.2
  Day 90, Type III, n=45, 24 | 13.3 | 8.3
  Day 90, Type IV, n=45, 24 | 13.3 | 12.5

4. Primary Outcome: Average Residual Lens Lysozyme
Description: Worn study lenses were removed and analyzed by high performance liquid chromatography (HPLC) for residual lens lysozyme (protein). Values reported as lower than the limit of quantitation or none detected were imputed as 0.5 μg or 0 μg, respectively. A lower value indicates less lysozyme deposition. One eye (study eye) contributed to the analysis.
Time Frame: Day 90/Early Exit
Population: This analysis population includes all randomized subjects.
Measure: Mean (Standard Deviation); unit: micrograms per lens
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 71 | 35
micrograms per lens | 0.2 (0.5) | 0.2 (0.4)

5. Primary Outcome: Percentage of Subjects With Change From Baseline in Contact Lens-Corrected Distance Visual Acuity (CLCDVA) by Line Change
Description: Distance VA was assessed for each eye individually while reading a chart distant to the participant in dimmed room illumination. VA was measured using a Snellen chart, with 20/20 Snellen acuity considered normal distance-eyesight. A line increase indicates an improvement in VA. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all subjects with data at visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 69 | 35
percentage of subjects
  Day 7, 2 Line Increase from Baseline | 0.0 | 0.0
  Day 7, 1 Line Increase from Baseline | 2.9 | 0.0
  Day 7, No Change from Baseline | 92.8 | 94.3
  Day 7, 1 Line Decrease from Baseline | 4.3 | 5.7
  Day 7, 2 Line Decrease from Baseline | 0.0 | 0.0
  Day 30, 2 Line Increase from Baseline | 0.0 | 0.0
  Day 30, 1 Line Increase from Baseline | 1.4 | 0.0
  Day 30, No Change from Baseline | 95.7 | 97.1
  Day 30, 1 Line Decrease from Baseline | 2.9 | 2.9
  Day 30, 2 Line Decrease from Baseline | 0.0 | 0.0
  Day 60, 2 Line Increase from Baseline | 1.4 | 0.0
  Day 60, 1 Line Increase from Baseline | 1.4 | 2.9
  Day 60, No Change from Baseline | 97.1 | 94.3
  Day 60, 1 Line Decrease from Baseline | 0.0 | 2.9
  Day 60, 2 Line Decrease from Baseline | 0.0 | 0.0
  Day 90, 2 Line Increase from Baseline | 0.0 | 2.9
  Day 90, 1 Line Increase from Baseline | 0.0 | 2.9
  Day 90, No Change from Baseline | 97.1 | 91.4
  Day 90, 1 Line Decrease from Baseline | 2.9 | 2.9
  Day 90, 2 Line Decrease from Baseline | 0.0 | 0.0

6. Primary Outcome: Average Lens Wear Time
Description: Subject recorded a response to the question, "Averaging over the last 3 days, how many hours per day did you wear your contact lenses?" Lens wear time was measured in hours.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all subjects with data at visit.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 69 | 35
Hours
  Day 7 | 12.3 (2.7) | 13.3 (2.4)
  Day 30 | 12.5 (2.7) | 12.7 (2.8)
  Day 60 | 11.8 (2.9) | 13.3 (2.6)
  Day 90 | 12.4 (2.8) | 13.1 (2.6)

7. Primary Outcome: Number of Unscheduled Lens Replacements by Reason
Description: No lens replacements were planned during the study. Lenses could be replaced as needed due to loss, damage, or as deemed necessary by the Investigator. If it became necessary to replace a lens, the subject was examined at an unscheduled visit. The counts in the table represent the total number of unscheduled lenses replaced by reason for any eye, any subject.
Time Frame: Up to Day 90
Population: This analysis population includes all randomized subjects.
Measure: Number; unit: lenses
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 71 | 35
lenses
  Lost | 3 | 1
  Lens torn on eye | 0 | 1
  Lens torn while handling | 1 | 0

8. Primary Outcome: Likert Item - "When I Use This Solution, my Lenses Are Comfortable All Day."
Description: Lens comfort was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all subjects with data at visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 69 | 35
percentage of subjects
  Day 7, Strongly Agree | 30.4 | 68.6
  Day 7, Agree | 52.2 | 28.6
  Day 7, Undecided | 7.2 | 0.0
  Day 7, Disagree | 10.1 | 2.9
  Day 7, Strongly Disgree | 0.0 | 0.0
  Day 30, Strongly Agree | 31.9 | 68.6
  Day 30, Agree | 47.8 | 28.6
  Day 30, Undecided | 4.3 | 2.9
  Day 30, Disagree | 13.0 | 0.0
  Day 30, Strongly Disagree | 2.9 | 0.0
  Day 60, Strongly Agree | 30.4 | 62.9
  Day 60, Agree | 49.3 | 28.6
  Day 60, Undecided | 8.7 | 0.0
  Day 60, Disagree | 10.1 | 5.7
  Day 60, Strongly Disagree | 1.4 | 2.9
  Day 90, Strongly Agree | 30.4 | 54.3
  Day 90, Agree | 50.7 | 28.6
  Day 90, Undecided | 1.4 | 2.9
  Day 90, Disagree | 15.9 | 11.4
  Day 90, Strongly Disagree | 1.4 | 2.9

9. Primary Outcome: Likert Item - "When I Use This Solution, at the End of the Lens Wearing Day my Vision is Clear."
Description: Clear vision was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all subjects with data at visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 69 | 35
percentage of subjects
  Day 7, Strongly Agree | 37.7 | 48.6
  Day 7, Agree | 40.6 | 45.7
  Day 7, Undecided | 2.9 | 0.0
  Day 7, Disagree | 15.9 | 5.7
  Day 7, Strongly Disagree | 2.9 | 0.0
  Day 30, Strongly Agree | 29.0 | 48.6
  Day 30, Agree | 53.6 | 45.7
  Day 30, Undecided | 7.2 | 2.9
  Day 30, Disagree | 10.1 | 2.9
  Day 30, Strongly Disagree | 0.0 | 0.0
  Day 60, Strongly Agree | 33.3 | 57.1
  Day 60, Agree | 49.3 | 28.6
  Day 60, Undecided | 4.3 | 5.7
  Day 60, Disagree | 11.6 | 8.6
  Day 60, Strongly Disagree | 1.4 | 0.0
  Day 90, Strongly Agree | 29.0 | 45.7
  Day 90, Agree | 49.3 | 34.3
  Day 90, Undecided | 7.2 | 5.7
  Day 90, Disagree | 13.0 | 14.3
  Day 90, Strongly Disagree | 1.4 | 0.0

10. Primary Outcome: Likert Item - "When I Use This Solution, I Like the Way This Product Feels During Handling."
Description: Product handling was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all subjects with data at visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 69 | 35
percentage of subjects
  Day 7, Strongly Agree | 23.2 | 48.6
  Day 7, Agree | 50.7 | 40.0
  Day 7, Undecided | 20.3 | 8.6
  Day 7, Disagree | 5.8 | 2.9
  Day 7, Strongly Disagree | 0.0 | 0.0
  Day 30, Strongly Agree | 26.1 | 57.1
  Day 30, Agree | 53.6 | 34.3
  Day 30, Undecided | 13.0 | 8.6
  Day 30, Disagree | 5.8 | 0.0
  Day 30, Strongly Disagree | 1.4 | 0.0
  Day 60, Strongly Agree | 26.1 | 51.4
  Day 60, Agree | 56.5 | 34.3
  Day 60, Undecided | 14.5 | 11.4
  Day 60, Disagree | 2.9 | 0.0
  Day 60, Strongly Disagree | 0.0 | 2.9
  Day 90, Strongly Agree | 27.5 | 48.6
  Day 90, Agree | 52.2 | 40.0
  Day 90, Undecided | 11.6 | 5.7
  Day 90, Disagree | 7.2 | 2.9
  Day 90, Strongly Disagree | 1.4 | 2.9

11. Primary Outcome: Crystalline Deposit Area Covered
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered. Values were reported as a percentage of lens area covered. One eye (study eye) contributed to the analysis.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of lens area
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 71 | 35
percentage of lens area
  Day 7, n=10, 5 | 18.0 (16.2) | 19.0 (18.2)
  Day 30, n=17, 3 | 13.6 (18.1) | 16.7 (20.2)
  Day 60, n=18, 8 | 11.9 (14.1) | 7.0 (3.5)
  Day 90, n=21, 10 | 18.1 (16.3) | 10.8 (14.5)

12. Primary Outcome: Film Deposit Area Covered
Description: as for outcome 11
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of lens area
Arm/Group | FID 120974A | Boston Simplus
Number analyzed (Participants) | 71 | 35
percentage of lens area
  Day 7, n=40, 15 | 23.8 (17.2) | 22.7 (13.7)
  Day 30, n=47, 20 | 26.2 (22.0) | 28.4 (21.1)
  Day 60, n=47, 20 | 26.4 (17.5) | 24.0 (11.0)
  Day 90, n=45, 24 | 25.3 (13.7) | 28.3 (21.9)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (Nov 2013 - May 2014). AEs were obtained as solicited and volunteered comments from subjects and as observations by the study Investigator as outlined in the study protocol.
Description: AEs were defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device or control product. AEs are reported as pre-treatment and treatment-emergent.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to exposure to investigational product
- FID 120974A: All subjects who were exposed to FID 120947A
- Boston Simplus: All subjects who were exposed to Boston Simplus
Arm/Group | Pre-treatment | FID 120974A | Boston Simplus
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/71 | 0/35
Other Adverse Events (participants affected / at risk) | 0/112 | 0/71 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.